CLINICAL TRIAL: NCT00729287
Title: Phase III Randomized Chemoprevention Study of Selenium on the Recurrence of Non-invasive Bladder Cancer
Brief Title: Selenium in Preventing Cancer Recurrence in Patients With Bladder Cancer
Acronym: SELEBLAT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: KU Leuven (Other)
Collaborators: Agentschap voor Innovatie door Wetenschap en Technologie (Other)
Responsible Party: Principal Investigator, Maria Goossens, Prof. dr. Frank Buntinx, KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CDR0000602239
Record Dates: First submitted 2008-08-06; First posted 2008-08-07 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Bladder Cancer
Keywords: stage 0 bladder cancer; stage I bladder cancer; transitional cell carcinoma of the bladder
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Selenium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Placebo Comparator): Patients receive oral placebo daily in addition to standard care.
  Interventions: Other: placebo
- Arm II (Experimental): Patients receive oral selenium daily in addition to standard care.
  Interventions: Dietary Supplement: selenium

INTERVENTIONS:
Dietary Supplement: selenium — Given orally
  Arms: Arm II
Other: placebo — Given orally
  Arms: Arm I

SUMMARY:
RATIONALE: Chemoprevention is the use of certain drugs to keep cancer from forming, growing, or coming back. The use of selenium may keep bladder cancer from growing or coming back. It is not yet known whether selenium is more effective than a placebo in preventing cancer recurrence in patients with bladder cancer.

PURPOSE: This randomized phase III trial is studying selenium to see how well it works compared with a placebo in preventing cancer recurrence in patients with bladder cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the effect of selenium, when administered with standard care, in preventing the recurrence of bladder cancer in patients with non-muscle-invasive transitional cell carcinoma of the bladder at risk for recurrence.

Secondary

* To determine the effect of selenium on the recurrence of bladder cancer, in terms of histological type, number, and size.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral placebo daily in addition to standard care.
* Arm II: Patients receive oral selenium daily in addition to standard care.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

Histopathologically confirmed non-muscle-invasive transitional cell carcinoma (TCC) of the bladder (< pT2 )

PATIENT CHARACTERISTICS:

* Able to swallow pills
* Not pregnant
* Fertile patients must use effective contraception
* No other malignancy within the past 5 years
* No known hypersensitivity or adverse reactions to selenium
* No other serious medical or psychiatric illness that would preclude giving informed consent
* No condition that, in the opinion of the investigator, may interfere with the safety of the patient or the evaluation of the study objectives

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* More than 30 days since prior daily dietary supplements containing selenium
* No other concurrent selenium (contained in individual supplements, antioxidant mix, or multivitamin) intake
* No concurrent participation in another study involving a medical, surgical, nutritional, or lifestyle intervention

  * Concurrent participation in the follow-up phase of another study allowed

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Actual)
Dates: Start 2009-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Effect of selenium in preventing the recurrence of bladder cancer | 3 years

SECONDARY OUTCOMES:
Effect of selenium on the progression of bladder cancer, in terms of histological type, number, and size | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Frank Buntinx, MD, PhD, Principal Investigator — Department of public Health, KU Leuven
Locations (1):
- Department of public Health, KU Leuven, Leuven, Belgium

REFERENCES:
- [Derived] Goossens ME, Buntinx F, Joniau S, Ackaert K, Ameye F, Billiet I, Braeckman J, Breugelmans A, Darras J, Dilen K, Goeman L, Kellen E, Tombal B, Van Bruwaene S, Van Cleyenbreuge B, Van der Aa F, Vekemans K, Van Poppel H, Zeegers MP. Designing the selenium and bladder cancer trial (SELEBLAT), a phase lll randomized chemoprevention study with selenium on recurrence of bladder cancer in Belgium. BMC Urol. 2012 Mar 21;12:8. doi: 10.1186/1471-2490-12-8. PMID 22436453